CLINICAL TRIAL: NCT06374069
Title: Longevity Families of the Netherlands
Acronym: LOF-NL
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Jacobijn Gussekloo, Prof. dr. (Unknown); Simon P. Mooijaart, Prof. dr. (Unknown)
Responsible Party: Principal Investigator, Eline Slagboom, Eline Slagboom, Prof. dr., Leiden University Medical Center
Other Study IDs: NL81887.058.23
Record Dates: First submitted 2024-03-20; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Longevity; Familial Longevity; Extreme Longevity; Aging

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases - Enriched for familial longevity: Siblings of dutch Caucasian descent ages 75 and older
- Controls - Non-enriched for familial longevity: Individuals of dutch Caucasian descent ages 75 and older solely in their family.

SUMMARY:
The demographic life expectancy enhancement of the past 150 years imposes an urgent challenge in Western and economically growing societies to stimulate the healthy lifespan that is lagging behind. Families surviving into exceptionally high ages (longevity) in good physical and mental health illustrate that this is physiologically possible. Such families harbor cross generational socio-genetic mechanisms that mediate healthy aging and protection from (multi)morbidity.

The purpose of our research is: to identify gene variants associated with healthy aging and protection from (multi)morbidity; to study the social-, environment- and behavioral factors of familial longevity, their role in (multi-)morbidity and its interaction with the genetic component.

ELIGIBILITY:
Inclusion Criteria:

* Siblings of Dutch Caucasian descent age 75+ enriched for familial longevity
* Individuals of Dutch Caucasian descent age 75+ who are not enriched for familial longevity

Exclusion Criteria:

-

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Dutch Caucasian descent:
  Ages 75 and older, with siblings enriched for familial longevity, and individuals without a history of familial longevity
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identifying the genetic variants of Familial Longevity | through study completion, an average of 2 years
  To identify gene variants associated with healthy aging and protection from (multi)morbidity

SECONDARY OUTCOMES:
Studying the environmental factor of Familial Longevity through questionnaires and its interaction with the genetic component | through study completion, an average of 2 years
  To study the social-, environment- and behavioral factors of familial longevity, their role in (multi-)morbidity and its interaction with the genetic component

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands